CLINICAL TRIAL: NCT02777255
Title: Evaluation of Genomic, Structural and Molecular Changes Associated With Severe Cardiac Allograft Vasculopathy in Heart Transplant Recipients
Brief Title: Severe CAV MRI in Heart Transplant Recipient
Status: Withdrawn | Type: Observational
Why Stopped: PI left University
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1103M96798
Record Dates: First submitted 2013-03-13; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Allograft Vasculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be saved in paxgene tubes for RNA sequencing
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: CAV is associated with fibrotic changes on cardiac MRI, altered levels of pathogenetically-related biomarkers, and specific RNA expression changes in the blood

DETAILED DESCRIPTION:
Cardiac allograft vasculopathy (CAV) is a major limitation to longevity after heart transplantation (HT), accounting for almost 30% of deaths after year 5. The only cure is re-transplant which is associated with a 30-day mortality of 30%, and raises ethical issues due to limited resources. Standard preventive measures, such as statin therapy, have limited success due to the multi-factorial nature of the process and influence of transplant-specific risk factors. Consensus regarding the management of CAV is lacking due to the absence of prospective studies evaluating timing of initiation of therapy, effect of therapies on long-term outcomes, and effective diagnostic strategies. Primary prevention of CAV, which will be evaluated in the proposed study, could improve longevity of heart transplant recipients and optimize use of a limited resource.

The current gold standard for evaluation of CAV is surveillance coronary angiogram, which is highly insensitive, particularly in early disease. Intravascular ultrasound (IVUS) is the most sensitive tool for the diagnosis of CAV, providing specific information such as the appearance and thickness of the intima and media, however it is not widely used in the clinical setting. Physiologic studies of the coronary arteries are also useful in assessing risk, but are not practical in a clinical setting. These invasive studies expose the heart transplant recipient to radiation, nephrotoxic contrast, and potential vascular complications. During the evolution of CAV, there are important structural, functional, and genomic changes that occur in parallel and possibly before.

Study Objectives

1. Determine the structural, functional and genomic changes associated with severe CAV
2. Identify novel and noninvasive markers of CAV

Study Design This is a cross-sectional study which will evaluate structural, functional and genomic changes associated with severe CAV in heart transplant recipients within 15 years of transplant. 30 heart transplant recipients identified via our study database and the transplant clinic will be enrolled into the study. We will enroll 15 heart transplant patients with severe CAV and 15 without CAV.

Subjects will undergo a one-time assessment of radial artery elasticity, blood draw for gene expression profiles, and cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Provide informed consent
* Successful orthotopic heart transplant within 15 years of enrollment

Exclusion Criteria:

* Chronic kidney disease with creatinine >2.5 mg/dl
* Ejection fraction <45% if CAV or <50% if no CAV
* IV contrast allergy or reaction (gadolinium)
* Active infection (febrile illness, cytomegalovirus or other significant infection)
* Treated humoral rejection or cellular rejection grade 3A/2R or greater within 3 months
* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplant patients with severe CAV and heart transplant patients without CAV
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline associated with severe CAV | 1 year
  Determine the structural (degree of fibrosis), functional and genomic changes associated with severe CAV

SECONDARY OUTCOMES:
Novel noninvasive markers of CAV from baseline | 1 year
  Identify novel and noninvasive markers of CAV

CONTACTS AND LOCATIONS:
Overall Officials: Monica M Colvin-Adams, MD.,MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States